CLINICAL TRIAL: NCT05931640
Title: Effects of Plyometric Training Versus Virtual Reality on Upper Limb Among Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of Plyometric Training Versus Virtual Reality Among Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0724
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hemiplegic cerebral palsy , virtual reality , plyometric training , upper limb
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual Reality Therapy that includes use of VR goggle, VR headset and play station if available. Virtual games like move-pro will be used for upper limb movements. A session of 12-45 minutes, twice weekly will be done. And scoring will be done with the help of additional tools.
  Interventions: Device: Virtual Reality
- Plyometric Training (Experimental): Plyometric therapy that includes 10 minutes of ball throwing, push-ups, jumping and hopping/skipping. At start intensity and speed is low, but will be increased gradually. Every score will be noted with the help of additional tools.
  Interventions: Device: Plyometric Training

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Therapy that includes use of VR goggle, VR headset and play station if available. Virtual games like move-pro will be used for upper limb movements. A session of 12-45 minutes, twice weekly will be done. And scoring will be done with the help of additional tools.
  Arms: Virtual Reality
Device: Plyometric Training — Plyometric therapy that includes 10 minutes of ball throwing, push-ups, jumping and hopping/skipping. At start intensity and speed is low, but will be increased gradually. Every score will be noted with the help of additional tools.
  Arms: Plyometric Training

SUMMARY:
The purpose of this study is to compare the effects of plyometric training versus virtual reality on upper limb among hemiplegic cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy is a combination of disorders that makes a child's life difficult; it mainly affects the motor abilities of the child. Cerebral palsy (CP) is a neurodevelopmental disorder characterized by abnormalities of muscle tone, movement and motor skills, and is attributed to injury to the developing brain. Children with cerebral palsy (CP) have decreased capacity to participate in play and sports activities. Reduced capacity to perform typical childhood activities contributes to low habitual physical activity and declining gross motor function in adolescence. Preceding more into this disorder there are 'hemiplegic cp'. Hemiplegic cp means that one side of the body is weak, paralyzed, it includes hand, arm, shoulder, leg of the affected side. For better treatments interventions are being invented day by day but according to my research.Plyometric therapy raises force and speeds your muscle contractions' force and speeds and strength training that leads to higher explosive power needed in sports and even everyday activities. Plyometric activities can be utilized in both the lower and upper extremities, with running, jumping, or throwing a ball and virtual reality therapy (use of virtual reality technology for psychological or occupational therapy and in affecting virtual rehabilitation.); which one is better for speedy recovery.

The tools used will be QUEST (Quality of Upper Extremity Skill Tests) and Ball & Box Test (BBT). Study will be conducted on 28 patients in two Groups. Group A will be Control Group that will be provided with Plyometric (push-ups, ball throwing, jumping, running, kicking). A protocol of 10 minutes of plyometric therapy will be given including running and jumping with ball throwing. and Group B will be Experimental Group that will be provided with Virtual Reality Therapy (VRT). A session of 12-45, twice a week, through VR goggles or VR will be given. QUEST and box & block test will be used as tools. The Control group will be administered with Plyometric therapy that includes 10 minutes of ball throwing, push-ups, jumping and hopping/skipping. At start intensity and speed is low, but will be increased gradually. Every score will be noted with the help of additional tools.The Experimental group will be administered with Virtual Reality Therapy that includes use of VR goggle, VR headset and play station if available. Virtual games like move-pro will be used for upper limb movements. A session of 12-45 minutes, twice weekly will be done. And scoring will be done with the help of additional tools.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 12 years.
* Lack of use of the affected upper limb.
* Level I-III of the Manual Ability Classification System (MACS).
* Students scoring of Modified Ashworth Scale should be 3 or less than 3 out of 5 for the same muscle groups.

Exclusion Criteria:

* Low cognitive level compatible with attending a special education
* school.
* Presence of contractures in the affected upper limb.
* Surgery in the six months previously.
* Botulinum toxin in the two months previously.
* Uncontrolled epilepsy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skill Tests | 4 weeks
  Quality of Upper Extremity Skills Test (QUEST) is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy
Ball & Box Test | 4 weeks
  The Box and Block Test (BBT) measures unilateral gross manual dexterity

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nosheen Manzoor, MS OPMT, Principal Investigator — Riphah International University
Locations (1):
- Govt. National special education centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No